CLINICAL TRIAL: NCT00648791
Title: Single-Dose Fasting In Vivo Bioequivalence Study of Finasteride Tablets (5 mg; Mylan) and Proscar Tablets (5 mg; Merck) in Healthy Male Volunteers
Brief Title: Fasting Study of Finasteride Tablets 5 mg and Proscar Tablets 5 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Will Sullvan, Global Head of Product Risk and Safety Management, Mylan Inc.
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: FINA-0460
Record Dates: First submitted 2008-03-30; First posted 2008-04-01 (Estimated); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Healthy
MeSH Terms: interventions — Finasteride

ARMS (2):
- 1 (Experimental): Finasteride Tablets 5 mg
  Interventions: Drug: Finasteride Tablets 5 mg
- 2 (Active Comparator): Proscar Tablets 5 mg
  Interventions: Drug: Proscar Tablets 5 mg

INTERVENTIONS:
Drug: Finasteride Tablets 5 mg — 5mg, single dose fasting
  Arms: 1
Drug: Proscar Tablets 5 mg — 5mg, single dose fasting
  Arms: 2

SUMMARY:
The objective of this study was to investigate the bioequivalence of Mylan's finasteride 5 mg tablets to Merck's Proscar® 5 mg tablets following a single, oral 5 mg (1 x 5 mg) dose administration under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years and older
2. Sex: Male During the course of the study, from study screen until study exit, male volunteers must use a spermicide-containing barrier method of contraception to prevent the pregnancy of their sexual partner. This advice should be documented in the informed consent form.
3. Weight: At least 60 kg (132 lbs) and all subjects within 15% of Ideal Body Weight (IBW), as referenced by the Table of "Desirable Weights of Adults" Metropolitan Life Insurance Company, 1999 (See Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
4. All subjects should be judged normal and healthy during a pre-study medical evaluation (physical examination, laboratory evaluation, Hepatitis B, Hepatitis C and HIV tests, 12-lead ECG, and urine drug screen including amphetamine, barbiturates, benzodiazepines, cannabinoid, cocaine, opiates, phencyclidine, and methadone) performed within 14 days of the initial dose of study medication.

Exclusion Criteria:

1. Institutionalized subjects will not be used.
2. Social Habits:

   1. Use of any tobacco products within one year prior to dosing.
   2. Ingestion of any alcoholic, caffeine- or xanthine-containing food or beverage within the 48 hours prior to the initial dose of study medication.
   3. Ingestion of any vitamins or herbal products within 7 days prior to the initial dose of the study medication.
   4. Any recent, significant change in dietary or exercise habits.
3. Medications:

   1. Use of any medication within the last 14 days prior to the initial dose of study medication, including over-the-counter medications.
   2. Use of any medication known to alter hepatic enzyme activity within 28 days prior to the initial dose of study medication.
4. Diseases:

   1. History of any significant chronic disease and/or hepatitis.
   2. History of drug and/or alcohol abuse.
   3. Acute illness at the time of either the pre-study medical evaluation or dosing.
   4. A positive HIV, Hepatitis B, or Hepatitis C test result.
5. Abnormal and clinically significant laboratory test results:

   1. Clinically significant deviation from the Guide to Clinically Relevant Abnormalities (See Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
   2. Abnormal and clinically relevant ECG tracing.
6. Donation or loss of a significant volume of blood or plasma (> 450 mL) within 28 days prior to the initial dose of study medication.
7. Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication.
8. Allergy or hypersensitivity to finasteride or other related products.
9. History of difficulties in swallowing, or any gastrointestinal disease which could affect the drug absorption.
10. Consumption of grapefruit or grapefruit containing products within 7 days of drug administration.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2004-09; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Dorian Williams, M.D., Principal Investigator — Kendle International Inc.
Locations (1):
- Kendle International Inc., Morgantown, West Virginia, United States

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html